CLINICAL TRIAL: NCT00376441
Title: Study of Sexual Function and Urinary Symptoms in Women Having Vaginal Surgeries
Brief Title: Evaluate Women After Vaginal Surgery for Urinary Symptoms and Sexual Function
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-119
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2011-08

CONDITIONS: Urinary Incontinence; Pelvic Organ Prolapse; Surgery
Keywords: vaginal; incontinence; sexual function
MeSH Terms: conditions — Urinary Incontinence; Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Vaginal Surgery — patients undergoing vaginal surgery

SUMMARY:
Assess the outcomes of vaginal surgeries and its impact on sexual function and urinary symptoms.

DETAILED DESCRIPTION:
Currently, up to 43% of women in the United States have female sexual dysfunction (FSD). In a recent study of 109 sexually active women in a urogynecology practice, FSD was noted using the validated Female Sexual Function Index (FSFI) in 64% of the women. Difficulties with sexual function are also associated with pelvic organ prolapse and urinary incontinence. One in nine women will have surgery for incontinence or prolapse in her lifetime. The impact of vaginal surgeries on sexual function and urinary symptoms has been scarcely reported in the literature. The methodology of most of those studies is flawed by the use of questionnaires that were not validated, small sample sizes and no comparison control group. In addition, several studies only focused on one surgical intervention, specific types of incontinence or prolapse, or both. It is difficult to make sense out of the discordant research findings when applying it to our patient population.

This is a prospective study of women with incontinence or pelvic organ prolapse. Subjects will be selected from three urology practices. All patients will be asked to complete a short patient history form. If the woman meets the study criteria, the study will be explained and if she agrees to participate in this study, informed consent will be obtained. She will then complete the FSFI, SF-12 and PFDI-20 questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years of age
* Having urinary incontinence or pelvic organ prolapse
* Capable of giving informed consent
* Capable and willing to follow all study related procedures

Exclusion Criteria:

* Reported history of urethral obstruction (not secondary to prolapse), stricture, bladder calculi or bladder tumor in the last 2 years.
* Pregnant as confirmed by urine pregnancy test or plans to become pregnant during the study period.
* Breast feeding
* Currently participating or have participated within the past 30 days in any clinical investigation involving or impacting urinary or renal function
* Cannot independently comprehend and complete the questionnaires.
* The subject is deemed unsuitable for enrollment in this study by the investigators based on their history or physical examination.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women at least 18 years of age having urinary incontinence or pelvic organ prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2006-08; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Peters, M.D., Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

REFERENCES:
- [Background] Norton P, Brubaker L. Urinary incontinence in women. Lancet. 2006 Jan 7;367(9504):57-67. doi: 10.1016/S0140-6736(06)67925-7. PMID 16399154
- [Background] Laumann EO, Paik A, Rosen RC. Sexual dysfunction in the United States: prevalence and predictors. JAMA. 1999 Feb 10;281(6):537-44. doi: 10.1001/jama.281.6.537. PMID 10022110
- [Background] Pauls RN, Segal JL, Silva WA, Kleeman SD, Karram MM. Sexual function in patients presenting to a urogynecology practice. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Nov;17(6):576-80. doi: 10.1007/s00192-006-0070-5. Epub 2006 Jun 8. PMID 16767528
- [Background] Weber AM, Walters MD, Schover LR, Mitchinson A. Sexual function in women with uterovaginal prolapse and urinary incontinence. Obstet Gynecol. 1995 Apr;85(4):483-7. doi: 10.1016/0029-7844(94)00434-F. PMID 7898820
- [Background] LeCroy C. Urinary incontinence occurring during intercourse: effect on sexual function in women. Urol Nurs. 2006 Feb;26(1):53-6. No abstract available. PMID 16562386